CLINICAL TRIAL: NCT03797820
Title: A Prospective, Multicenter,Registry Study of Aortic Valve Stenosis in Zhejiang Elderly
Brief Title: Multicenter Registry Study of Aortic Valve Stenosis in Zhejiang Elderly（Mrs AVS）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Jinhua Central Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); The Central Hospital of Lishui City (Other); Sir Run Run Shaw Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZJU CT012
Record Dates: First submitted 2018-12-24; First posted 2019-01-09 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Our study type is observational — Our study type is observational

SUMMARY:
Aortic valve stenosis (AVS) is becoming more and more frequent with the aging, which has brought a heavy burden to the world. However, the prevalence and prognosis of valvular heart disease are not so clear, especially in the developing countries such as China etc. Because of the slow and progressive nature of AVS, symptoms might not be too severe to be diagnosed on time. Our retrospective survey (Int J Cardiol. 2016 Nov 25) indicated that severe aortic valve stenosis are very common in China. Hence, we design a prospective, observational cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective ,treatments and prognosis of Chinese elderly patients with aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 60 years old meet the following condition moderate or above aortic stenosis as defined by echocardiography: Aortic stenosis, moderate or above, or valve area≤1.5cm2, or maximal jet velocity ≥3.0m/sec, or mean pressure gradient≥20mmHg

Exclusion Criteria:

1. Patients cannot be followed up for any reasons.
2. Patients in critical condition may be die in one year.
3. Patients have been enrolled in this study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years old and moderate or above aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality,disabling strokes and Surgical or transcatheter aortic valve replacement | one year
  time from enrolled to first occurrence of any of the components of the composite outcome

SECONDARY OUTCOMES:
Hospitalization for heart failure | one year
  time from enrolled to first occurrence of the outcome
Surgical or transcatheter aortic valve replacement | one year
  time from enrolled to first occurrence of the outcome
Cardiovascular death | one year
  time from enrolled to first occurrence of the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Hu P, Liu XB, Liang J, Zhu QF, Pu CX, Tang MY, Wang JA. A hospital-based survey of patients with severe valvular heart disease in China. Int J Cardiol. 2017 Mar 15;231:244-247. doi: 10.1016/j.ijcard.2016.11.301. Epub 2016 Nov 25. PMID 27908608
- See also: A hospital-based survey of patients with severe valvular heart disease in China — http://www.ncbi.nlm.nih.gov/pubmed/27908608